CLINICAL TRIAL: NCT00695383
Title: Early Exercise in Critically Ill Patients Enhances Short-Term Functional Recovery
Brief Title: Early Exercise Training in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Prof. Dr. Rik Gosselink, Department of Rehabilitation Sciences, Katholieke Universiteit Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G 0523.06
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Critical Illness; Intensive Care; Muscle Weakness; Deconditioning
Keywords: Exercise therapy; Physiotherapy; Critical illness; Intensive care; Muscle weakness; Mechanical ventilation
MeSH Terms: conditions — Critical Illness; Muscle Weakness | interventions — Exercise Therapy; Exercise; Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Bedside cycle exercise therapy
- 2 (Active Comparator)
  Interventions: Behavioral: Standard physiotherapy program

INTERVENTIONS:
Behavioral: Bedside cycle exercise therapy — A 20-minute cycling exercise session is performed 5 days a week using a bedside cycle ergometer. Patients can cycle passively and actively against increasing resistance. Besides this, patients receive the standard physiotherapy program as in arm 2
  Other Names: exercise therapy; exercise training; exercise; cycle training; cycle exercise; Motomed Letto
  Arms: 1
Behavioral: Standard physiotherapy program — The standard physiotherapy program consists of daily chest physiotherapy and a mobilization session on 5 days per week.
  Other Names: Usual physiotherapy; Routine physiotherapy; Mobilization
  Arms: 2

SUMMARY:
This randomized controlled trial was designed to investigate whether a daily training session using a bedside cycle ergometer, started early in stable critically ill patients with an expected prolonged ICU stay, could induce a beneficial effect on exercise performance, quadriceps force and functional autonomy at ICU and hospital discharge compared to a standard physiotherapy program.

DETAILED DESCRIPTION:
Inactivity during prolonged bed rest leads to muscle dysfunction. Muscle function decreases even faster in ICU patients due to inflammation, pharmacological agents (corticosteroids, muscle relaxants, neuromuscular blockers, antibiotics), and the presence of neuromuscular syndromes, associated with critical illness. A recent recommendation document advices to start early with active and passive exercise in critically ill patients. However, no evidence is available concerning the feasibility of an early muscle training intervention in the acute ICU phase when patients are still under sedation. A rather new method to train bed-bound patients is the use of a bedside cycle ergometer. This randomized controlled trial was designed to investigate whether a daily training session using a bedside cycle ergometer, started early in stable critically ill patients with an expected prolonged ICU stay, could induce a beneficial effect on exercise performance, quadriceps force and functional autonomy at ICU and hospital discharge compared to a standard physiotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* ICU stay > 5 days
* Expected prolonged stay of at least 7 more days
* Cardiorespiratory status that allows at least passive exercise therapy

Exclusion Criteria:

* Persistent or progressive neurological or (neuro)muscular disease
* Coagulation disorders (INR > 1.5, [BP] < 50000/mm³)
* Intracranial pressure > 20 mmHg
* Psychiatric disorders or severe confusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
six-minute walking distance | hospital discharge

SECONDARY OUTCOMES:
quadriceps force | ICU discharge and hospital discharge
functional status (Berg Balance Scale, Functional Ambulation Categories, SF-36 Physical Function-item) | ICU discharge and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rik Gosselink, PT, phD, Study Director — Department of Rehabilitation Sciences, University Hospitals KULeuven; Chris Burtin, PT, MSc, Principal Investigator — Department of Rehabilitation Sciences, University Hospitals KULeuven
Locations (1):
- Department of Rehabilitation Sciences, University Hospitals KULeuven, Leuven, Vlaams-Brabant, Belgium